CLINICAL TRIAL: NCT06711380
Title: Patient Ambassador in Gynecologic Oncology Clinical Trials
Brief Title: Patient Ambassador
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Emily Ko, MD, Medical Director, Pennsylvania Hospital Abramson Cancer Center, Director, Gynecologic Oncology Populations Sciences Research Program, Director, REACH - Research Equity Center for Gynecologic Cancers and Health, Abramson Cancer Center at Penn Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UPCC 33823; 854317 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2024-10-18; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Gynecologic Cancer
Keywords: mentor; ambassador; gynecologic cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer Ambassador (Other): There is one arm of the trial which includes the Patient Ambassador intervention.
  Interventions: Other: Peer Ambassador

INTERVENTIONS:
Other: Peer Ambassador — Patient mentor (patient with history of gynecologic cancer who has experience with clinical trials) one on one discussion with patient mentee (patient receiving standard of care treatment for gynecologic cancers).

SUMMARY:
The overall objective of this study is to design and evaluate a peer ambassador intervention to improve gynecologic cancer trial enrollment. The primary Aim is to determine the possibility of using peer ambassadors to increase discussion, awareness, and enrollment of patients with advanced or recurrent gynecologic cancer onto clinical trials.

DETAILED DESCRIPTION:
Participants will participate in a peer ambassador program where a patient ambassador (mentor) will be paired with a mentee. The patient ambassador will be a patient with history of gynecologic cancer who has experience with clinical trials and can serve as an ambassador to facilitate discussions regarding education and awareness of clinical trials. This discussion will potentially assist mentees to make informed decisions about their engagement in discussing clinical trials, looking for clinical trials, and desire and acceptance of clinical trials. This will also allow ambassadors to gain information about perceived barriers regarding clinical trials.

The investigators seek to identify patient ambassadors, who will be trained to lead 1:1 discussion with patient mentees. Each ambassador will be paired with up to 5 mentees. Each ambassador-mentee pairing will have 1-2 encounters (meetings) over the course of 12 months. The total number of encounters and the total number of ambassador-mentee dyads created, will be logged.

Enrollment and study visits will occur over a 12 month period. Each mentor will be in the study approximately one year, and each mentee will be in the study approximately 2 months.

ELIGIBILITY:
Mentee Inclusion Criteria:

* Eligible subjects will include those with advanced gynecologic cancer (metastatic or persistent/progressive disease despite primary treatment) or high-risk gynecologic cancer undergoing active systemic therapy not currently enrolled on clinical trials. These patients include those starting a new line of chemotherapy, or who have a diagnosis needing chemotherapy.
* Patients will be identified from the UPHS gynecologic oncology and medical oncology clinics serving gynecologic cancer patients (Penn Medicine Washington Square, PCAM/HUP, Radnor, Chester County, Penn Medicine Cherry Hill). Clinic rosters over 6 months intervals will be screened for eligibility.
* Patients who have been discussed at tumor board conferences and recommended to consider clinical trials will screened for recruitment.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the ambassador program | 12 months
  Feasibility of the ambassador program will be assessed using the Feasibility of Intervention Measure (FIM). The FIM is a 4-item questionnaire measuring the feasibility of an intervention.
Acceptability of the ambassador program | 12 months
  Acceptability of this program will be assessed using AIM (Acceptability of Intervention Measure). The AIM is a 4-item questionnaire measuring the acceptability of an intervention.
Intention | 12 months
  Intention to recommend the ambassador program will be assessed using the Net Promoter Score (NPS) measure. NPS instrument is attached in the appendix and does not require any licensing agreement for use in this research study. Participants will be asked to rate the likelihood of their referral of the program on a scale of zero to ten (zero to six is a "Detractor", while scores of seven to eight are "Passives" and scores of nine and ten are "Promoters").

SECONDARY OUTCOMES:
Mentee knowledge | 2 months
  Mentee knowledge regarding clinical trials before and after their discussion session(s) with ambassador. This will be assessed using a knowledge of clinical trials questionnaire.
Sociodemographic | 2 months
  Sociodemographic and clinical factors associated with feasibility, acceptability, and likelihood to recommend this program.
Clinical trial enrollment | 12 months
  Proportion of mentees in this program who enrolled onto a clinical trial

CONTACTS AND LOCATIONS:
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will share data arising from the proposed project to the extent that it is permissible and consistent with the prevailing data use agreements and controlling IRBs. Data sharing will occur in a timely fashion. Following acceptance for publication of the main findings from the final data set, the investigators will provide for the timely release and sharing of the de-identified data from the cohort study and the qualitative interviews. These data sets will be provided upon written request to all interested investigators. Upon acceptance for publication of the main study findings, the investigators will also share upon written request with interested investigators the code used in analyzing data.